CLINICAL TRIAL: NCT05629533
Title: The Nanowear Wearable System SimpleSense Validation Trial for Cardiac Output, Cardiac Power Output and Pulmonary Artery Pressure.in Patients Undergoing Right Heart Catheterization
Brief Title: The Nanowear Wearable System SimpleSense Validation Trial for Cardiac Output
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanowear Inc. (Industry)
Collaborators: Westchester Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0044
Record Dates: First submitted 2022-11-10; First posted 2022-11-29 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Right Heart Catheterization
Keywords: Cardiac output; Right heart catheterization; SimpleSense; Algorithm; Pulmonary Artery Pressure; Heart failure; Endomyocardial biopsy; Cardiogenic shock
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Phase 1: Subjects to undergo right heart catheterization SimpleSense data collected from the first set of subjects and associate the data from SimpleSense to the right heart catheterization values.
  Undergoing right heart catheterization for a clinical indication including but not limited to :
  * Prognosis of advanced heart failure
  * During endomyocardial biopsy
  * Candidacy for heart transplant
  * Management of cardiogenic shock
  Interventions: Device: SimpleSense
- Phase 2: Subjects to undergo right heart catheterization SimpleSense data collected from the second set of subjects and evaluate the algorithms developed to estimate cardiac output from SimpleSense data. The second set of subjects are from within the sample population that are sequestered from the first set used for association of data from SimpleSense to the data from the right heart catheterization.
  Interventions: Device: SimpleSense

INTERVENTIONS:
Device: SimpleSense — The study is observational only. No interventions will be triggered by the SimpleSense device

SUMMARY:
The Nanowear SimpleSense study is a single center, prospective, non-randomized, feasibility, non- significant risk study The study will be done in 2 phases. Phase 1 will use SimpleSense data collected from the first set of subjects and associate the data from SimpleSense to the right heart catheterization values.' Phase 2 will evaluate the algorithms developed to estimate cardiac output from SimpleSense data using a second set of subjects from within the sample population that are sequestered from the first set used for association of data from SimpleSense to the data from the right heart catheterization.

DETAILED DESCRIPTION:
Patients undergoing right heart catheterization for a clinical indication including but not limited to prognosis for advanced heart failure, during endomyocardial biopsy, candidacy for heart transplant or management of cardiogenic shock.

Study Design:

The Nanowear SimpleSense study is a single center, prospective, non-randomized, feasibility, non- significant risk study The study will be done in 2 phases. Phase 1 will use SimpleSense data collected from the first set of subjects and associate the data from SimpleSense to the right heart catheterization values.' Phase 2 will evaluate the algorithms developed to estimate cardiac output from SimpleSense data using a second set of subjects from within the sample population that are sequestered from the first set used for association of data from SimpleSense to the data from the right heart catheterization.

Number of subjects and sites:

The Nanowear SimpleSense study will enroll up to 100 subjects to collect data at Westchester Medical Center. The testing will include a SimpleSense device recording and simultaneous measurement of Cardiac Output, and Pulmonary Artery Pressure by right heart catheterization.

Duration of study:

The duration of the Nanowear SimpleSense study is expected to be 1 year.

Study Population:

Subjects of legal age to give informed consent who are undergoing right heart catheterization for a clinical indication including but not limited to :

* Prognosis of advanced heart failure
* During endomyocardial biopsy
* Candidacy for heart transplant
* Management of cardiogenic shock

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent
2. Male or female over the age of 18 years
3. The patient is undergoing right heart catheterization

Exclusion Criteria:

1. Subject unwilling or unable to comply with wearing the Nanowear SimpleSense System.
2. Subjects who are pregnant
3. Severe aortic stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of legal age to give informed consent who are
  Undergoing right heart catheterization for a clinical indication including but not limited to :
  * Prognosis of advanced heart failure
  * During endomyocardial biopsy
  * Candidacy for heart transplant
  * Management of cardiogenic shock
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac output algorithm | 9-12 months
  To establish a correlation between the SimpleSense and the cardiac output from the right heart catheterization.
Algorithm for Pulmonary Artery Pressure | 9 -12 months
  To train a model for Pulmonary Artery Pressure estimation based on the data acquired for SimpleSense against the Pulmonary Artery Pressure data from the right heart catheterization
Algorithm for Pulmonary Wedge Pressure | 9-12 months
  To train a model for Pulmonary Wedge Pressure estimation based on the data acquired for SimpleSense against the Pulmonary Wedge Pressure data from the right heart catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Westchester Medical Center, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No